CLINICAL TRIAL: NCT01119144
Title: Comparing the Reconstruction of the Orbit Fracture With a Poly Caprolactone / Tri-Calcium Phosphate ( PCL/TCP ) Implant vs. a Titanium Mesh Implant.
Brief Title: Polycaprolactone / Tricalcium Phosphate (PCL/TCP) v Titanium Orbital Implant : Randomised Trial
Acronym: PCL/TCP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: LIM THIAM CHYE / Professor, National University Hospital / National Unviersity of Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NUHS/SUR/2010/1; D / 08 / 465 (Registry Identifier: D / 08 / 465)
Record Dates: First submitted 2010-05-05; First posted 2010-05-07 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-04

CONDITIONS: Fractures; Enophthalmos; Diplopia
Keywords: Orbital; fractures; enophthalmos; diplopia; eye
MeSH Terms: conditions — Fractures, Bone; Enophthalmos; Diplopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Polycaprolactone / Tricalcium Phosphate (Experimental): Polycaprolactone / Tricalcium Phosphate group to assess efficacy of new implant
  Interventions: Device: Polycaprolactone / Tri-Calcium Phosphate
- Control (Active Comparator): Control group with titanium mesh
  Interventions: Device: Titanium Mesh

INTERVENTIONS:
Device: Polycaprolactone / Tri-Calcium Phosphate — Orbital implant for reconstruction of the orbital walls
  Other Names: Osteomesh Tri-Calcium Phosphate (TCP)
  Arms: Polycaprolactone / Tricalcium Phosphate
Device: Titanium Mesh — Titanium mesh for comparison to Polycaprolactone / Tri-Calcium Phosphate (PCL / TCP) mesh
  Other Names: Titanium Orbital mesh
  Arms: Control

SUMMARY:
Hypothesis: Polycaprolactone / Tricalcium Phosphate Orbital (PCL / TCP) Implant is as effective in the reconstruction of the Orbital walls as Titanium Mesh implant.

In this study we will be conducting a randomised trial to compare implants made of 2 materials for Orbital reconstruction

* Polycaprolactone / Tricalcium Phosphate (PCL / TCP)
* Titanium

Patients to be recruited :

* 80 randomised equally into the 2 groups
* age range: 21 - 70
* includes orbital wall defects from trauma, after osteotomies
* excludes patients with Diabetes Mellitus, known allergies to polycaprolactone & its analogues, know allergies to Tricalcium Phosphate & its analogues, infections generalised & around the orbital region

Trial Duration: April 2010 - March 2015

Follow up:

* postoperative 1 week, 1 month, 3 months, 6 months, and 12 months
* Computer Tomographic (CT) scan of Orbits immediate postoperative and at 12 months appointment

DETAILED DESCRIPTION:
Hypothesis: Polycaprolactone / Tricalcium Phosphate (PCL / TCP) Orbital Implant is as effective in the reconstruction of the Orbital walls as Titanium Mesh

In this study we will be conducting a randomised trial to compare implants made of 2 materials for Orbital reconstruction

* Polycaprolactone / Tricalcium Phosphate (PCL / TCP)
* Titanium

Patients to be recruited :

* 80 randomised equally into the 2 groups
* age range: 21 -70
* includes orbital wall defects from trauma confirmed by Computer Tomographic (CT) scans, after osteotomies
* excludes patients with Diabetes Mellitus, known allergies to polycaprolactone & its analogues, know allergies to Tricalcium Phosphate & its analogues, infections generalised & around the orbital region

Trial Duration : April 2010 - March 2015

Follow up:

* postoperative 1 week, 1 month, 3 months, 6 months, and 12 months
* Computer Tomographic (CT) scan of Orbits immediate postoperative and at 12 months appointment
* all patients will be seen & assessed in the Plastic & Ophthalmology outpatient clinics by Principal Investigator (PI) and collaborators

End point :

* endpoint for follow-up is 12 months
* all patients are assessed for assessed for diplopia, enophthalmos, exophthalmos, visual acuity, mobility of the globe, contour symmetry
* all patients will have a Computer Tomographic (CT) scan of the orbits at 12 months to assess the bony orbit & orbital volume
* patients will be discharged from follow up at 12 months if asymptomatic
* patients with complications will exit the protocol & will be treated on their merits eg. infection - removal of implant, etc

Data Management :

* maintained by the Principal Investigator (PI) under repository of the Research & Development Office, National Healthcare Group (NHG) / National University Health Systems (NUHS), Singapore
* no data will be released without the permission of the Principal Investigator (PI) & the Research & Development Office, National Healthcare Group (NHG) / National University Health Systems (NUHS), Singapore

ELIGIBILITY:
Inclusion Criteria:

* age 21 y - 70 y
* both males / females included
* orbital fractures
* defect after orbital osteotomies

Exclusion Criteria:

* patient refusal
* infection around the orbit / generalised infection
* Diabetes mellitus
* allergies to polycaprolactone & its analogues
* allergies to titanium

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-04; Primary Completion 2015-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Enophthalmos | 1 year
  Assess the presence of enophthalmos after reconstruction of the orbital walls at 1 week, 1 month, 3 months, 6 months and 12 months

SECONDARY OUTCOMES:
Diplopia | 1 year
  Assess the evidence of diplopia on follow up at 1 week, 1 month, 3 months, 6 months and 12 months
motility of the globe | 1 year
  assess globe motility on follow up at 1 week, 1 month, 3 months, 6 months, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Thiam Chye Lim, MD, Principal Investigator — Natioanl University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore